CLINICAL TRIAL: NCT05442411
Title: Regional Scalp Block Versus IV Parecoxib for Post-operative Cranioplasty Surgery Pain: A Comparison of Pain Score.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Mohamad Hasyizan Hassan, Senior Lecturer and Neuroanaesthesiologist, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USM/ JEPeM/19080504
Record Dates: First submitted 2022-06-28; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; parecoxib

STUDY DESIGN:
Intervention Model Description: randomised contrrolled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: participant is blineded to the treatment as they was givemn intraopeartively the pain score assessor is blinded since the assessment was done postoperatively
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- post operative pain score (Experimental): post operative pain score at 1hour, 2 hour, 4 hour, 6 hour, and 12 hour
  Interventions: Drug: Ropivacaine 0.75% Injectable Solution
- morphine requirement (Experimental): post operative PCA morphine requirement
  Interventions: Drug: Ropivacaine 0.75% Injectable Solution

INTERVENTIONS:
Drug: Ropivacaine 0.75% Injectable Solution — comparison of scalp block vs conventional post operative parecoxib
  Other Names: parecoxib 40mg

SUMMARY:
To compare the post cranioplasty pain score using scalp block versus conventional analgesia using IV Parecoxib and requirement of morphine between two groups as rescue analgesia

DETAILED DESCRIPTION:
This study involved a prospective, double-blinded randomized controlled trial which has been approved by the Medical Research and Ethics Committee (JEPEM) of Universiti Sains Malaysia (JEPeM Code: USM/ JEPeM/19100637).

Fifty-eight patients with written informed consent and American Society of Anaesthesiologist (ASA) physical status I and II, aged 18 to 60 years old, pre-operative GCS of 15 and underwent elective cranioplasty surgery under general anaesthesia (GA) between September 2019 until March 2022 were selected for the study and randomized by computer generated randomization into two groups; Regional Scalp Block (n = 29) and IV Parecoxib (n = 29). The patients were excluded from this study if they were a known allergy to local anesthesia or NSAIDS, had risk for bleeding tendency or coagulopathy, low preoperative platelets count (< 100 x103/mL) or with underlying bronchial asthma. The patient withdrawn from the study if he or she was not able to score post pain using Visual analog Scale (VAS) or had redo surgery for postoperative bleeding.

During surgery, all of them were induced by standard anaesthesia protocol. They were given IV fentanyl 1-2mcg/kg, IV propofol 2 mg/kg and IV rocuronium 0.6mg /kg. The anaesthesia was maintained with sevoflurane with minimum alveolar concentration (MAC) of 1.0 to 1.2 with mixture of air and oxygen. The intraoperative analgesia were IV Fentanyl 1-2mcg/kg and IV paracetamol 1g. The total intraoperative analgesia dose was recorded in GA form and the top-up muscle relaxant was given as needed upon evidence of rebreathing in the capnograph waveform. At the end of the surgery, all subjects were reversed with IV neostigmine 0.05 mg/kg and atropine 0.02mg/kg.

The injection solution for both groups were prepared by the single anaesthesiologist who are experience and familiar with scalp block procedure and IV Parecoxib. For the Group A, they were given regional scalp block by using solution 0.375% ropivacaine and lidocaine 1% up to 20 ml. The same person was performed the Scalp Block by injecting the solution into Supra-orbital & Supratrochlear (V1), Auriculo-temporal (V2), Post-auricular branches of the Greater Auricular Nerves and Occipital nerves after the surgeon completed skin closure of the scalp at the end of surgery (at the side that will be operated). Group B was injected IV parecoxib 40mg during the closure of the scalp. All subjects will be reversed using standard reversal and fulfil criteria for extubation before extubation Post cranioplasty operation, both groups were given PCA Morphine as rescue analgesia if pain score ≥ 4. Both groups received IV paracetamol 1g 6 hourly as additional analgesia.

Pain score was assessed by staff nurses in the ward (unrelated to study to avoid bias) by using visual analogue scale (VAS) at interval hours of first, second, forth, sixth and twelfth-hour post cranioplasty. The patient was withdrawn from the study if they had massive bleeding or hemodynamically unstable or require intensive care and ventilatory support post cranioplasty. The patients and post-operative assessors (the staff nurse in the ward) were blind to avoid bias.

After 12 hours, the total requirement of morphine and time for request rescue analgesia were recorded. The side effects of both methods were documented. Local anesthesia side effects such as allergic reactions, local tissue, cardiovascular, central nervous system, and systemic toxicity, infection, changes in wound healing, or increased wound drainage. Parecoxib side effects such as bleeding, renal failure, and myocardial infarction.

The sample size was calculated using the G*Power Software (Version 3.1.9.7 by Franz Faul, Universitat Keil, Germany. Based on the objective to compare effectiveness in pain control between both groups using effect size f 0.30, power of 0.8, ɑ error probability 0.05, number of groups 2 and number of measurements 5. It required 21 peoples in one group and a total sample size of 42. These included a 10% dropout.

Data were analysed using IBM SPSS statistics version 26 software. All measurement data were analysed for normal distribution and homogeneity variance. All demographic data between groups were analysed using descriptive analysis and independent sample t-test for numerical data and Chi-square analysis for categorical data. Differences in pain score using VAS between two groups were analysed using one-way and two-way repeated ANOVA. Model assumptions of normality and homogeneity of covariance were checked. Total morphine requirement and the first time PCA were analysed using an independent sample t-test. The side effects of both groups were analysed using the Chi-Square test. A P -the value of < 0.05 was regarded as statistically significant.

ELIGIBILITY:
Fifty-eight patients with written informed consent and American Society of Anaesthesiologist (ASA) physical status I and II, aged 18 to 60 years old, pre-operative GCS of 15 and underwent elective cranioplasty surgery under general anaesthesia (GA) between September 2019 until March 2022 were selected for the study and randomized by computer generated randomization into two groups; Regional Scalp Block (n = 29) and IV Parecoxib (n = 29). The patients were excluded from this study if they were a known allergy to local anesthesia or NSAIDS, had risk for bleeding tendency or coagulopathy, low preoperative platelets count (< 100 x103/mL) or with underlying bronchial asthma. The patient withdrawn from the study if he or she was not able to score post pain using Visual analog Scale (VAS) or had redo surgery for postoperative bleeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
pain score | 12 hours
  visual analog score

SECONDARY OUTCOMES:
total morpine requirement | 12 hours
  PCA post operatively

CONTACTS AND LOCATIONS:
Locations (1):
- School Of Medical Sciences, Health Campus, Universioti Sains Malaysia, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided
further study in the process